CLINICAL TRIAL: NCT02552680
Title: Influence of a Preventive Program (Educational and Gymnastics) for Work-Related Musculoskeletal Disorders in Surgeons
Brief Title: Preventive Program for Work-Related Musculoskeletal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GPPG100432
Record Dates: First submitted 2015-08-18; First posted 2015-09-17 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Quality of Life
Keywords: Work-Related Musculoskeletal Disorders; Quality of life; Health Education
MeSH Terms: conditions — Health Education | interventions — Exercise; Guidelines as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise + guideline (Experimental): Participants will participate in eight meetings consisting of exercise and guidelines on care and prevention of Work-Related Musculoskeletal Disorders in activities of daily living, especially those relating work activities.
  Interventions: Other: Exercise; Other: Guideline
- brochure (Active Comparator): Participants will receive a manual-brochure - containing information about general health.
  Interventions: Other: Brochure

INTERVENTIONS:
Other: Exercise — Physical Exercise
  Arms: Exercise + guideline
Other: Guideline — Guideline on care and prevention of Work-Related Musculoskeletal Disorders in activities of daily living, especially those relating work activities.
  Arms: Exercise + guideline
Other: Brochure — Manual/brochure containing information about general health
  Arms: brochure

SUMMARY:
Introduction: Work-Related Musculoskeletal Disorders (WMSDs) are characterized by inflammation of muscles, tendons, fascia and nerves of upper limbs, shoulder girdle and neck. Its incidence is increasing and there is evidence of its association with the pace of work. As WMSDs, another major public health problem is back pain, which also negatively influence the quality of life of patients. These diseases affect many workers, among them, workers in the health area, including surgeons. Studies show that many surgeons are suffering from fatigue and musculoskeletal pain after undergoing surgery, especially laparoscopy. Regarding the quality of life of doctors, a study indicates that surgeons have commitment of domains "Vitality" and "Pain". For these reasons it is important to develop strategies for prevention of occupational risks (WMSDs) in this class of workers.

Objectives: To evaluate the influence of a Preventive Program (educational and gymnastics) for prevention of WMSDs, in the quality of life, in limitation of the work, in intensity and frequency of musculoskeletal pain in surgeons of the Hospital de Clínicas de Porto Alegre. There will also be evaluated the effects of the program on muscular strength and flexibility of medics participating in the Preventive Program.

Methodology: Randomized clinical trial with a sample of 54 surgeons, divided into two groups: A ("Intervention": will participate in eight meetings consisting of exercise and guidelines on care and prevention of WMSDs in activities of daily living, especially those relating work activities) and B ("Control": will receive a manual-brochure - containing information about general health). Participants will sign a Letter of Consent.

DETAILED DESCRIPTION:
Clinical Trial Study with 54 surgeons allocated in two groups: A and B. They received two protocols in accordance with the groups they have been allocated.

Group A: participated in eight meetings supervised by physical education professionals, with 15 minutes duration, individually administered, twice a week, during the surgeons working hours, at times and places combined with them. The meetings were composed of endurance exercise, mobility and muscle stretching. They were also given guidance on care and prevention of Work-Related Musculoskeletal Disorders in activities fo daily life, especially those related to work activities.

Group B: received a manual (brochure ) containing information on general health care, especially designed for this study. With food guide, sleep, physical activity and smoking.

Were measured the quality of life, muscle force, muscle stretching and pain. The dates were collected at the beginning of the procedures, 4 weeks after the protocols and 26 after the protocols.

ELIGIBILITY:
Inclusion Criteria:

* surgeons (teachers, contractors and medical residents)
* of the Hospital de Clínicas de Porto Alegre
* members of General Surgery teams, Digestive Surgery , Plastic Surgery and Coloproctology
* of both sexes

Exclusion Criteria:

* individuals who did not agree to participate in the study
* those who were not present at the time of the study (regardless of reason)
* those who had some more serious illness that prevented the achievement of study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | 26 weeks after the interventions
  Quality of life evaluated by the Short-Form Survey Questionnaire (SF-36). Unit of measure: Scale of Quality of life.

SECONDARY OUTCOMES:
Muscle strength - Grip and Pinch Strength | 4 weeks and 26 weeks after the interventions
  Evaluated by hand grip dynamometer and pinch grip dynamometer. Unit of measure: kilogram force (kgf) (both evaluations).
Muscle flexibility | 4 weeks and 26 weeks after the interventions
  Evaluated by "Banco de Wells". Unit of measure: centimeters (cm)
Musculoskeletal intensity of pain | 4 weeks and 26 weeks after the interventions
  Evaluated by Questionnaire. Unit of measure: Scale of pain.
Quality of life - after 4 weeks | 4 weeks after the interventions
  Quality of life evaluated by the Short-Form Survey Questionnaire (SF-36). Unit of measure: Scale of Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Antônio C dos Santos, Doctorate, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided